CLINICAL TRIAL: NCT02511054
Title: Sanaria PfSPZ Challenge With Pyrimethamine Chemoprophylaxis (PfSPZ-CVac Approach): Phase 1 Trial to Determine Safety and Protective Efficacy of Sanaria PfSPZ Challenge With Concurrent Pyrimethamine Treatment That Inhibits Development of Asexual Blood Stages of Plasmodium Falciparumc
Brief Title: Sanaria PfSPZ Challenge With Pyrimethamine Chemoprophylaxis (PfSPZ-CVac Approach): Phase 1 Trial to Determine Safety and Protective Efficacy of Sanaria PfSPZ Challenge With Concurrent Pyrimethamine Treatment That Inhibits Development of Asexual B...
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150169; 15-I-0169
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06-01

CONDITIONS: Malaria
Keywords: Immunogenicity; Liver Stage; Parasites; Blood; Infection
MeSH Terms: conditions — Malaria; Infections | interventions — Chloroquine; Pyrimethamine

ARMS (4):
- 1a (Experimental): Arm 1a (n=2), the pilot phase, is designed to examinethat the dosing of PYR on 2, 3 days post DVI with Sanaria PfSPZ Challenge while under CQ prophylaxis does not result in subpatent parasitemia (positive qRT-PCR result defined as two consecutive samples > 20 parasites/uL or a single positive qRTPCR (Bullet) 100) or a single episode of patent parasitemia (positive blood smear defined as two unambiguous parasites in a thicksmear) in (Bullet)1/2 subjects. Subjects will considered enrolled into the study upon receipt of the loading dose of CQ (2 days prior to administration of first dose of Sanaria PfSPZ Challenge).
  Interventions: Drug: Chloroquine (CQ); Drug: Pyrimethamine (PYR); Biological: Sanaria PfSPZ Challenge (NF54)
- 2 (Experimental): Arm 2 (n=12) will receive the selected regimen of pyrimethamine, on 2, 3 days (unless another Arm other than Arm 1a is determined from the pilot phase) post Sanaria PfSPZ Challenge via DVI while under CQprophylaxis. These subjects will be considered enrolledinto the study upon receipt of the loading dose of CQ(2 days prior to administration of first dose of Sanaria PfSPZ Challenge).
  Interventions: Drug: Chloroquine (CQ); Drug: Pyrimethamine (PYR); Biological: Sanaria PfSPZ Challenge (NF54)
- 3 (Experimental): Arm 3 (n=6) will receive Sanaria PfSPZ Challenge DVI while under CQ prophylaxis without PYR treatment. These subjects will be considered enrolled into the study upon receipt of the loading dose of CQ (2 days prior to administration of first dose of Sanaria PfSPZ Challenge).
  Interventions: Drug: Chloroquine (CQ); Biological: Sanaria PfSPZ Challenge (NF54)
- 4 (Experimental): Arm 4 (n=5) will only receive one dose of Sanaria PfSPZ Challenge at CHMI as a positive control for thestudy. Subjects in Arm 4 will be considered enrolledon the day of Sanaria PfSPZ Challenge via DVI.
  Interventions: Biological: Sanaria PfSPZ Challenge (NF54)

INTERVENTIONS:
Drug: Chloroquine (CQ) — Chloroquine Phosphate is a 4-aminoquinoline compound that is commercially available for oral administration. It is a white, odorless, bitter tasting, crystalline substance freely soluble in water; and widely used for the treatment andprophylaxis of malaria. It is supplied and manufactured in tablets of 500 mg (equivalent to 300 mg chloroquine phosphaste base)
  Arms: 1a; 2; 3
Drug: Pyrimethamine (PYR) — PYR is a folic acid antagonist that is commercially available; and has been commonly used as antimalarial drug for both treatment and prevention of malaria, usually in combination with sulfadoxine in adults, pregnant women, and children worldwide. It is manufactured in tablets of 25 mg.
  Arms: 1a; 2
Biological: Sanaria PfSPZ Challenge (NF54) — Sanaria PfSPZ Challenge are aseptic, cryopreserved P.falciparum sporozoites used for CHMI trials, produced by the biotechnology company; Sanaria Inc. In brief, manufacture includes the production, under traditional environmental conditions, of eggs from a colony of A. stephensi mosquitoes housed in a controlled environmental chamber. The sporozoites are purified, counted, and, at a specified concentration, cryopreserved. Cryopreservation commences with the addition of cryoprotective additives to the purified sporozoites to produce the Sanaria PfSPZ Challenge product. Sanaria PfSPZ Challenge is dispensed into screw-cap vials containing 15,000, 50,000, or 100,000 PfSPZ in a 20 L aliquot. Sanaria PfSPZ Challenge is stored in liquid nitrogen vapour phase at 140 (Infinite)C to -196 (Infinite)C.

SUMMARY:
Background:

- Malaria is a severe infection caused by a parasite. People can get malaria if a mosquito that carries the parasite bites them. Although malaria does not occur in the United States, many people in Africa, Asia, and South America do get malaria. In some cases, malaria can cause death. In 2013 alone, 584,000 people died due to malaria. Researchers want to find ways to prevent and treat malaria.

Objective:

- To find out if combining live, infectious malaria parasites (known as Sanaria PfSPZ Challenge) and two FDA approved drugs that kill malaria parasites (pyrimethamine [PYR] and chloroquine [CQ]) is safe and can provide people protection against malaria. The Sanaria PfSPZ Challenge has been used in other studies without significant side effects.

Eligibility:

* Healthy people ages 18-50 who weigh less than 170 pounds and are not pregnant or breastfeeding
* No history of hepatitis B, hepatitis C, or HIV infection
* Not currently enrolled in a clinical trial that involves a research drug or vaccine
* Have not traveled to an area with high malaria transmission within the last 5 years
* Never diagnosed with malaria in the past

Design:

* Participants will be in 1 of 4 groups.
* Participants will receive a combination of injections and drugs. What combination they will receive will depend on what group they are in. This combination of injections and drugs may include:

  * Injections of Sanaria PfSPZ Challenge (live, infectious malaria parasites) into a vein
  * FDA approved antimalarial drug called chloroquine (CQ)
  * FDA approved antimalarial drug called pyrimethamine (PYR)
  * FDA approved antimalarial drug called Malarone
  * The study will last approximately 3-7 months (depending on which group participants are in).
* There will be up to 68 study visits for three groups. One group will have up to 27 study visits. During the study visits, participants may have:

  * Medical history review
  * Physical exams
  * Electrocardiogram (ECG): soft electrodes will be placed on the skin. A machine will record the heart s electrical signals to evaluate heart function.
  * Blood and urine tests
  * Medication given in the clinic under direct observation
  * Injection of Sanaria PfSPZ Challenge into a vein
  * Participants will receive a diary, thermometer, and ruler to record their body temperature and any symptoms.

DETAILED DESCRIPTION:
Human studies have shown that immunization by the bite PfSPZ-infected mosquitoes under drug coverage with chloroquine, an approach called chemoprophylaxis with sporozoites (CPS), infection treatment vaccination (ITV), or chemoprophylaxis vaccination (CVac) can provide high level, long term protection against homologous controlled human malaria infection (CHMI). The Sanaria PfSPZ-CVac approach duplicates this with an injectable sporozoite (SPZ) regimen (aseptic, purified, cryopreserved SPZ). In both approaches, whether mosquitoes or a syringe are used for SPZ administration, when chloroquine is used as the chemoprophylactic agent, transient, limited, asexual erythrocytic stage (AES) parasitemia develops. However, exposure to liver stage parasites only, without having any parasites completing liver stage development and entering the blood, thereby reducing the potential to induce blood stage immunity, likewise has been shown in animal studies to induce protective immunity upon subsequent challenge with homologous parasites, indicating that the transient parasitemia is not integral to inducing protection. To achieve this requires a different partner drug regimen that includes activity against liver stage parasites.

Our approach, using PfSPZ-CVac with pyrimethamine (PYR), will assess this in humans. This phase 1 study will investigate the safety, tolerability, immunogenicity, and protective efficacy following liver stage only parasite exposure of direct venous inoculation (DVI) with aseptic, purified, cryopreserved Plasmodium falciparum (Pf) sporozoites (Sanaria PfSPZ Challenge), under chloroquine and pyrimethamine chemoprophylaxis, to induce stage specific sterile protection. By adding pyrimethamine chemoprophylaxis to chloroquine, liver stages will develop but should be killed before merozoites are released into the blood stream. The subjects will thus be exposed only to liver stage parasites (qPCR and blood smear negative). With this strategy, we will determine if protective immunity can develop without exposure to AES parasites and additionally whether it will minimize clinical symptoms associated with blood stage exposure. The timing of the pyrimethamine dose is critical to ensure the efficacy of pyrimethamine as causal prophylaxis, yet still allow for maximal antigenic exposure of liver-stage parasites to the host. An additional potential benefit of preventing AES parasitemia is the elimination of the immunosuppression associated with AES parasitemia.

This trial will be the first step in establishing a new regimen for the PfSPZ-CVac approach, exposure to liver stage parasites without subsequent blood stage parasites, assessing protection against homologous CHMI. In future trials, the two-drug regimen can be assessed for protection against heterologous Pf infection and longevity of protection. The results of the study will contribute to understanding the targets and mechanisms of immunity against Pf malaria infection.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a subject to participate in this trial:

1. Age greater than or equal to 18 and less than or equal to 50 years.
2. In good general health and without clinically significant medical history
3. Malaria comprehension exam completed, passed (a score of greater than or equal to 80% or per investigator s discretion) and reviewed prior to enrollment
4. Reliable access to the clinical trial center and availability to participate for duration of study
5. Females of childbearing potential must be willing to use reliable contraception (as defined below) from 21 days prior to study day -2 to 28 days following last Sanaria .

   * Subject to the judgment and discretion of the PI, female participants who meet ANY ONE of the criteria listed immediately below, may not be required to take any additional measures to avoid pregnancy. Such participants will be counseled on risks at the time of consent and at appropriate points (e.g. when pregnancy testing occurs) during the study:

     * Females who have had their uterus, and/or BOTH ovaries removed
     * Females who have had BOTH fallopian tubes surgically tied or removed
     * Females who are above the age of 45 and have spontaneously had no menses at any point during the past 12 or more consecutive months (i.e. have reached menopause)
     * Females who, in the conservative and reasonable judgment of the PI (e.g. due to sexual orientation or serious life choice (such as being celibate clergy or transgender), during the entire trial will NOT participate in any potentially reproductive sexual contact
     * Females who, in the conservative and reasonable judgment of the PI, are in a monogamous stable relationship with a male who has undergone vasectomy at least 4 months prior or another procedure/medical condition that deems the male sterile
   * Subject to the judgment and discretion of the PI, female participants who DO NOT meet ANY of the criteria listed above, will be appropriately counseled on reproductive risks and pregnancy avoidance, and will be required to adhere to the following measures and agree to 2 methods of pregnancy prevention as noted below:

CATEGORY 1:

* a highly effective hormonal method to prevent pregnancy [e.g. CONSISTENT, CONTINUOUS use of contraceptive pill, patch, ring, implant or injection], and/or
* IUD or equivalent

IN ADDITION TO

CATEGORY 2:

-a barrier method to be used at the time of potentially reproductive sexual activity (e.g. [male/female condom, 'cap,' or diaphragm] plus spermicide).

EXCLUSION CRITERIA:

A subject will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Currently is breast-feeding (if female).
2. Pregnancy as determined by a positive urine or serum human choriogonadotropin (beta-hCG) test at any point during the study (if female).
3. Recent travel to a malaria endemic area within 5 years of enrollment
4. Planned travel to a malaria endemic area during the study period
5. History of confirmed malaria diagnosis on peripheral blood smear or by clinical history in the past 10 years.
6. Hemoglobin, WBC, platelets, ALT, and creatinine outside of local lab normal range (subjects may be included at the investigator s discretion for not clinically significant values outside of normal range)
7. Abnormal urinalysis as defined by positive urine glucose, protein, and hemoglobin. Subject can be included if investigator determine the abnormality is not clinically significant .
8. Anticipated use during the study period, or use within the following periods prior to enrollment:

   1. Investigational malaria vaccine within the last five years
   2. Malaria chemoprophylaxis within 6 months
   3. Chronic systemic immunosuppressive medications (>14 days) within 6 months (e.g.cytotoxic medications, oral/parental corticosteroids >0.5 mg/kg/day prednisone or equivalent). Corticosteroid nasal spray for allergic rhinitis and topical corticosteroids for mild, uncomplicated dermatitis are allowed.
   4. Blood products or immunoglobulins within 6 months
   5. Systemic antibiotics with antimalarial effects within 30 days (such as clindamycin, doxycycline)
   6. Investigational or non-registered product or vaccine within 30 days
   7. Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to Sanaria PfSPZ Challenge
   8. Medications known to interact with pyrimethamine, chloroquine, atovaquone, proguanil (during the study period only)
9. History of:

   1. Sickle cell disease, sickle cell trait, or other hemoglobinopathies
   2. Splenectomy or functional asplenia
   3. Systemic anaphylaxis
   4. Any allergic reactions to study drugs
   5. Documented history of chronic or active neurologic disease (including seizures, uncontrolled migraine headaches)
   6. Psoriasis or porphyria
   7. Ocular diseases including retinopathy or visual field defects
10. Clinically significant medical condition, physical examination findings, other clinically

    significant abnormal laboratory results, or past medical history that may have clinically significant implications for current health status and participation in the study in the opinion of the Investigator. A clinically significant condition or process includes but is not limited to:
    1. A process that would affect the immune response, or requires medication that affects the immune response
    2. Any contraindication to repeated phlebotomy
    3. A condition or process in which signs or symptoms could be confused with reactions to malaria challenge and/or infection, including dermatologic abnormalities at the site of sporozoite inoculation
    4. A chronic or subclinical condition which could be exacerbated by administration of any of the PfSPZ-CVac components or malaria infection
11. Weight > 77.2 Kg at the time of screening (this will result in a minimum dose of pyrimethamine of approximately 0.7mg/Kg for a 50mg daily dose). (Note not required for Arm 4 CHMI controls)
12. History of, or known active cardiac disease including: (1) prior myocardial infarction (heart attack); (2) angina pectoris; (3) congestive heart failure; (4) valvular heart disease; (5) cardiomyopathy; (6) pericarditis; (7) stroke or transient ischemic attack; (8) exertional chest pain or shortness of breath; or ( 9) other heart conditions under the care of a doctor
13. Clinically significant ECG findings, as determined by the expert study cardiologist
14. Moderate or high risk for coronary heart disease (CHD) based on NHANES I cardiovascular risk assessment
15. Acute illness at the time of enrollment
16. Infection with HIV, Hepatitis B, Hepatitis C
17. Psychiatric condition that precludes compliance with the protocol including but not limited to:

    1. Psychosis within the past 3 years
    2. Ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
18. Suspected or known current alcohol or drug abuse as defined by the American Psychiatric Association in the DSM V at the discretion of the PI
19. Clinical trial staff and/or Sanaria employees with direct involvement in the conduct of the trial are excluded from participation.
20. Participating in other clinical trials involving investigational interventions or off label medication use during the study period (excluding participation in the optional long term follow up visits). Participation in other trials such as observational or imaging studies will be discussed with the investigators.
21. Any other finding that, in the judgment of the Investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a subject s ability to give informed consent, or increase the risk of having an adverse outcome from participating in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-07-21; Primary Completion 2016-10-21 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of local and systemic adverse events (AEs) and serious adverse events (SAEs) occurring after each Sanaria PfSPZ Challenge (Safety) | Approximately 6 months
(Pilot Phase Only) P. falciparum blood stage infection defined as detection of P. falciparum parasites by sensitive research qRT-PCR following Sanaria PfSPZ Challenge during first CVac regimen (Prevention of Pf Infection) | Approximately 3 months

SECONDARY OUTCOMES:
P. falciparum blood stage infection defined as detection of at least 2 P.falciparum parasites by microscopic examination of 0.5 L of blood or two consecutive positive diagnostic qRTPCR following homologous CHMI. (Protective Efficacy) | Approximately 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Healy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203
- [Background] Bijker EM, Bastiaens GJ, Teirlinck AC, van Gemert GJ, Graumans W, van de Vegte-Bolmer M, Siebelink-Stoter R, Arens T, Teelen K, Nahrendorf W, Remarque EJ, Roeffen W, Jansens A, Zimmerman D, Vos M, van Schaijk BC, Wiersma J, van der Ven AJ, de Mast Q, van Lieshout L, Verweij JJ, Hermsen CC, Scholzen A, Sauerwein RW. Protection against malaria after immunization by chloroquine prophylaxis and sporozoites is mediated by preerythrocytic immunity. Proc Natl Acad Sci U S A. 2013 May 7;110(19):7862-7. doi: 10.1073/pnas.1220360110. Epub 2013 Apr 18. PMID 23599283
- [Background] Sheehy SH, Spencer AJ, Douglas AD, Sim BK, Longley RJ, Edwards NJ, Poulton ID, Kimani D, Williams AR, Anagnostou NA, Roberts R, Kerridge S, Voysey M, James ER, Billingsley PF, Gunasekera A, Lawrie AM, Hoffman SL, Hill AV. Optimising Controlled Human Malaria Infection Studies Using Cryopreserved P. falciparum Parasites Administered by Needle and Syringe. PLoS One. 2013 Jun 18;8(6):e65960. doi: 10.1371/journal.pone.0065960. Print 2013. PMID 23823332
- [Derived] Mwakingwe-Omari A, Healy SA, Lane J, Cook DM, Kalhori S, Wyatt C, Kolluri A, Marte-Salcedo O, Imeru A, Nason M, Ding LK, Decederfelt H, Duan J, Neal J, Raiten J, Lee G, Hume JCC, Jeon JE, Ikpeama I, Kc N, Chakravarty S, Murshedkar T, Church LWP, Manoj A, Gunasekera A, Anderson C, Murphy SC, March S, Bhatia SN, James ER, Billingsley PF, Sim BKL, Richie TL, Zaidi I, Hoffman SL, Duffy PE. Two chemoattenuated PfSPZ malaria vaccines induce sterile hepatic immunity. Nature. 2021 Jul;595(7866):289-294. doi: 10.1038/s41586-021-03684-z. Epub 2021 Jun 30. PMID 34194041